CLINICAL TRIAL: NCT03957174
Title: Noradrenaline, Acetylcholine and Dynamic Learning in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R62807/RE001
Record Dates: First submitted 2019-05-10; First posted 2019-05-21 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — Reboxetine; Rivastigmine

STUDY DESIGN:
Intervention Model Description: Three group parallel design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Overencapsulated drug/placebo capsule used. Investigator and participant blind to allocation. Randomisation schedule drawn up by independent researcher and kept in locked cabinet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reboxetine (Experimental): Single dose of 4mg
  Interventions: Drug: Reboxetine
- Rivastigmine (Experimental): Single dose of 3mg
  Interventions: Drug: Rivastigmine
- Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Reboxetine — Single dose used to increase central norepinepherine
  Arms: Reboxetine
Drug: Rivastigmine — Single dose to increase central acetylcholine
  Arms: Rivastigmine
Drug: Placebo oral tablet — Single dose as control condition
  Arms: Placebo

SUMMARY:
The aim of this study is to characterize the role of central norepinephrine and acetylcholine on reward and emotion related information processing in healthy volunteers using behavioural tasks and pupillometry (with eye tracking equipment). The pharmacological compounds used in the study (reboxetine and rivastigmine) are used as tools to manipulate these systems rather than to treat patients. The aim of the study is not to study the clinical effects, pharmacodynamics, adverse reactions, absorption, distribution, metabolism or excretion of the drugs. Further, the population studied is non-clinical, the drugs are not administered in a therapeutic dosing regimen (only a single dose of study drug will be administered) and the investigators do not measure clinically significant outcomes.

DETAILED DESCRIPTION:
Background: Previous research has shown that human learners are able to encode the probabilities of positive and negative outcomes in parallel, and adjust their learning behaviour to the information content of positive and negative outcomes (Pulcu and Browning 2017). In reinforcement learning tasks, the volatility (also known as unexpected uncertainty arising when the environment changes suddenly) of outcomes directly influences how informative the outcomes are perceived to be (Behrens, Woolrich et al. 2007). Previous studies consistently shown that human participants use a higher learning rate while learning from outcomes with high volatility (Behrens, Woolrich et al. 2007, Browning, Behrens et al. 2015, Pulcu and Browning 2017). Another source of uncertainty is expected uncertainty, which arises from naturally varying outcomes (e.g. day to day changes in temperature). Different sources of uncertainty in the environment are argued to be associated with the activity of different neurotransmitter systems in the human brain (Yu and Dayan, 2005)(Angela and Dayan 2005). For example, outcome volatility (unexpected uncertainty) is thought to be associated with the activity of the central norepinephrine (NE) system, whereas outcome variation (expected uncertainty) has been linked to the cholinergic (ACY) system.

Studies using pupillometry (a non-invasive way of inferring central norepinephrine activity in the human brain) showed that pupil size is associated with the volatility of outcomes during reinforcement learning tasks (Browning, Behrens et al. 2015, Pulcu and Browning 2017). However, pupil size can also be influenced by the activity of other neurotransmitters including acetylcholine limiting the degree to which these results can be attributed to the NE system. Further, previous human studies have been associational in nature and thus the causal role of the NE and ACY systems in human learning under uncertainty have yet to be tested. The current study will address this knowledge gap by investigating how administering a single dose of the norepinephrine reuptake inhibitor reboxetine or cholinesterase inhibitor rivastigmine influence choice behaviour and pupillary correlates of human reinforcement learning.

Study Structure: All participants will be recruited via the recruitment pipeline described below. The randomisation procedure used will treat participants as if 2 parallel studies were running: a reboxetine vs. placebo and a rivastigmine vs. placebo study. Researchers will assign participants to either the reboxetine or rivastigmine arm (NB researchers will not be blind to this allocation although participants will be). Both studies will randomise participants in a 1:1 ratio, stratified by gender, to either the active drug or placebo (NB both researchers and participants will remain blind to this allocation). This will result in an overall group size for the reboxetine:rivastigmine:placebo groups of 30:30:60 (with participants randomised to placebo being specifically associated with the reboxetine or rivastigmine group). The rationale for this approach is that, while study procedures are identical for all participants, the investigators are addressing 2 separate questions in this study (the effect of NE manipulation and the effect of ACY manipulation on learning) which are more straightforwardly assessed using two, separate, placebo controlled comparisons rather than a larger three group study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age: 18 to 45 years
* Good physical and mental health
* Participant is willing and able to give informed consent for participation in the study
* Sufficient knowledge of English language to understand and complete study tasks
* Willingness to refrain from driving, cycling, or operating heavy machinery on the day of the study

Exclusion Criteria:

* Current or past psychiatric disorder (e.g. depression, bipolar disorder etc.)
* BMI outside of range 187.5 and 2530
* Any severe medical condition not stabilized at the time of the experiment that, in the opinion of the study medic, would compromise the safety or conduct of the study including significant hypertension (diastolic pressure > 100mmHg) or bradycardia (pulse less than 50 bpm).
* Any history of seizures, glaucoma or pancreatitis
* Lactose intolerance
* Any current or past physical illness that has the potential to significantly affect mental functioning (e.g. epilepsy, hypothyroidism, Parkinson's disease, multiple sclerosis etc.)
* Pregnant, or lactating woman
* Sexually active woman who does not use any medically accepted method of contraception
* Current or previous intake (last month) of any medication that has a significant potential to affect mental functioning (e.g. benzodiazepines, antidepressants, neuroleptics etc.)
* Any intake of recreational drugs in the last 3 months (e.g. marijuana, ecstasy etc.)
* Harmful alcohol use in the last 6 months (harmful alcohol use established based on self-reported work-related or social problems due to alcohol use or other's feedback to the participant that s/he should cut down)
* History of allergic reactions to relevant substances (reboxetine, rivastigmine)
* Previous participation in a study using the same or similar tasks
* In the researcher's or study medic's opinion participation in the study could be harmful or severely distressing to the participant (e.g. intolerance of side effects) or the participant is not able to follow instructions or complete study tasks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in learning rates | 2 hours after dosing (NB outcome is the change from the baseline measure to this time point)
  Learning rates from negative and positive outcomes received in a reinforcement learning task

SECONDARY OUTCOMES:
Pupil size | 2 hours after dosing (NB outcome is the change from the baseline measure to this time point)
  High temporal resolution pupil size measurement during a reinforcement learning task
Affective processing | 2 hours after dose
  Response accuracy in the Facial Emotion Recognition Task (FERT).

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Psychiatry, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Annonymised data and study protocol will be made available to researchers who contact the PI
Supporting Information: Study Protocol, Analytic Code
Time Frame: After completion of data analysis, and then indefinitely.
Access Criteria: Researchers who contact the PI with a valid interest in the data (as assessed by the PI)